CLINICAL TRIAL: NCT00989391
Title: A Double Blind (3rd Party Open), Randomized, Placebo Controlled, Dose Escalation Study To Investigate The Safety, Toleration, And Pharmacokinetics Of Multiple Oral Doses Of PF-03654764 In Healthy Subjects
Brief Title: A Study In Healthy People To Investigate The Safety, Toleration And Time Course Of Blood Concentrations Of Multiple Doses Of PF-03654764, Given By Mouth
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B0711002
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-12

CONDITIONS: Healthy
Keywords: Phase 1 multiple dose safety toleration pharmacokinetic
MeSH Terms: interventions — 3-fluoro-3-(3-fluoro-4-(pyrrolidin-1-ylmethyl)phenyl)-N-(2-methylpropyl)cyclobutanecarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Subjects will be assigned to receive either PF-03654764 or placebo.
  Interventions: Drug: PF-03654764; Drug: placebo
- Cohort 2 (Experimental): Subjects will be assigned to receive either PF-03654764 or placebo.
  Interventions: Drug: PF-03654764; Drug: placebo
- Cohort 3 (Experimental): Subjects will be assigned to receive either PF-03654764 or placebo.
  Interventions: Drug: PF-03654764; Drug: placebo

INTERVENTIONS:
Drug: PF-03654764 — 5mg orally once daily for 10 days. After satisfactory review of the available safety, toleration and PK data, progression to the next dose will occur if the last dose was well tolerated. If the previous dose was not well tolerated, after review of the safety data, and discussion between the Pfizer Study Team and the Investigator, the same dose may be given again, a lower dose within the tolerated dose range may be given, or the study may be stopped. The dose increments will be based on emerging safety and toleration data, as well as plasma exposure estimates and forward predictions of PK. Nominal administered doses will not exceed 24 mg per day.
  Arms: Cohort 1
Drug: placebo — orally once daily for 10 days. After satisfactory review of the available safety, toleration and PK data, progression to the next dose will occur if the last dose was well tolerated. If the previous dose was not well tolerated, after review of the safety data, and discussion between the Pfizer Study Team and the Investigator, the same dose may be given again, a lower dose within the tolerated dose range may be given, or the study may be stopped. The dose increments will be based on emerging safety and toleration data, as well as plasma exposure estimates and forward predictions of PK. Nominal administered doses will not exceed 24 mg per day.
  Arms: Cohort 1
Drug: PF-03654764 — 12mg orally once daily for 10 days. After satisfactory review of the available safety, toleration and PK data, progression to the next dose will occur if the last dose was well tolerated. If the previous dose was not well tolerated, after review of the safety data, and discussion between the Pfizer Study Team and the Investigator, the same dose may be given again, a lower dose within the tolerated dose range may be given, or the study may be stopped. The dose increments will be based on emerging safety and toleration data, as well as plasma exposure estimates and forward predictions of PK. Nominal administered doses will not exceed 24 mg per day.
  Arms: Cohort 2
Drug: placebo — orally once daily for 10 days. After satisfactory review of the available safety, toleration and PK data, progression to the next dose will occur if the last dose was well tolerated. If the previous dose was not well tolerated, after review of the safety data, and discussion between the Pfizer Study Team and the Investigator, the same dose may be given again, a lower dose within the tolerated dose range may be given, or the study may be stopped. The dose increments will be based on emerging safety and toleration data, as well as plasma exposure estimates and forward predictions of PK. Nominal administered doses will not exceed 24 mg per day.
  Arms: Cohort 2
Drug: PF-03654764 — 12mg orally twice daily on Days 1-9, and once on Day 10 After satisfactory review of the available safety, toleration and PK data, progression to the next dose will occur if the last dose was well tolerated. If the previous dose was not well tolerated, after review of the safety data, and discussion between the Pfizer Study Team and the Investigator, the same dose may be given again, a lower dose within the tolerated dose range may be given, or the study may be stopped. The dose increments will be based on emerging safety and toleration data, as well as plasma exposure estimates and forward predictions of PK. Nominal administered doses will not exceed 24 mg per day.
  Arms: Cohort 3
Drug: placebo — oral twice daily on Days 1-9 and once on Day 10. After satisfactory review of the available safety, toleration and PK data, progression to the next dose will occur if the last dose was well tolerated. If the previous dose was not well tolerated, after review of the safety data, and discussion between the Pfizer Study Team and the Investigator, the same dose may be given again, a lower dose within the tolerated dose range may be given, or the study may be stopped. The dose increments will be based on emerging safety and toleration data, as well as plasma exposure estimates and forward predictions of PK. Nominal administered doses will not exceed 24 mg per day.
  Arms: Cohort 3

SUMMARY:
The purpose of this study in heathy people is to investigate the safety, toleration and time course of PF-03654764 in the blood, following multiple doses given once or twice daily by mouth for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
safety & toleration: Adverse events, vital signs, 12 lead ECG, blood and urine safety tests, suicidality assessment using the Suicidality Tracking Scale (STS) and physical examination. | 10 days

SECONDARY OUTCOMES:
Plasma pharmacokinetics: Cmax, Tmax, AUCtau, t½, AUCtau (Day 10)/AUCtau (Day 1), CL/F | 10 days
Urine pharmacokinetics: Ae24 & Ae24% (for once daily doses) or Ae12 & Ae12% (for twice daily dose) on Day 10, CLR | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore